CLINICAL TRIAL: NCT01397825
Title: A Multicenter, Phase 1-2 Study of MLN8237, an Oral Aurora A Kinase Inhibitor, in Patients With Relapsed or Refractory Aggressive B-Cell Lymphoma Treated With Rituximab and Vincristine
Brief Title: MLN8237 in Patients With Relapsed or Refractory Aggressive B-Cell Lymphoma Treated With Rituximab +/- Vincristine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C14011; 2011-000609-32 (EudraCT Number); U1111-1181-0333 (Registry Identifier: WHO); 12/NE/0268 (Registry Identifier: NRES)
Record Dates: First submitted 2011-07-17; First posted 2011-07-20 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Diffuse Large B-Cell Lymphoma; Transformed Follicular Lymphoma; Mantle Cell Lymphoma; Burkitt's Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Burkitt Lymphoma | interventions — MLN 8237; Rituximab; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Safety Lead-in (Experimental): Alisertib 50 mg, enteric coated tablets (ECT), orally, twice daily (BID), on Days 1 to 7 followed by a 14-day rest period in 21-day cycles plus rituximab 375 mg/m^2, intravenous (IV), infusion on Day 1 of each 21-day cycle for up to 8 cycles. Following 8 cycles of treatment (or early discontinuation of rituximab) all participants with documented disease response or stabilization may continue with alisertib single-agent therapy for up to 2 years.
  Interventions: Drug: Alisertib (MLN8237); Drug: Rituximab
- Dose Escalation, Alisertib 30 mg (Experimental): Alisertib 30 mg, ECT, orally, BID, on Days 1 to 7 followed by a 14-day rest period plus rituximab 375 mg/m^2, IV, infusion on Day 1, plus vincristine 1.4 mg/m^2 (max 2 mg), IV, on Days 1 and 8 in a 21-day cycle for up to 8 cycles. Following 8 cycles of treatment (or early discontinuation of rituximab and/ or vincristine) all participants with documented disease response or stabilization may continue with alisertib single-agent therapy for up to 2 years.
  Interventions: Drug: Alisertib (MLN8237); Drug: Rituximab; Drug: Vincristine
- Dose Escalation, Alisertib 40 mg (Experimental): Alisertib 40 mg, ECT, orally, BID, on Days 1 to 7 followed by a 14-day rest period plus rituximab 375 mg/m^2, IV, infusion on Day 1 plus vincristine 1.4 mg/m^2, IV (max 2mg), on Days 1 and 8 in a 21-day cycle for up to 8 cycles. Following 8 cycles of treatment (or early discontinuation of rituximab and/ or vincristine) all participants with documented disease response or stabilization may continue with alisertib single-agent therapy for up to 2 years.
  Interventions: Drug: Alisertib (MLN8237); Drug: Rituximab; Drug: Vincristine
- Dose Escalation, Alisertib 50 mg (Experimental): Alisertib 50 mg, ECT, orally, BID, on Days 1 to 7 followed by a 14-day rest period plus rituximab 375 mg/m^2, IV, infusion on Day 1 plus vincristine 1.4 mg/m^2, IV (max 2mg), on Days 1 and 8 in a 21-day cycle for up to 8 cycles. Following 8 cycles of treatment (or early discontinuation of rituximab and/ or vincristine) all participants with documented disease response or stabilization may continue with alisertib single-agent therapy for up to 2 years.
  Interventions: Drug: Alisertib (MLN8237); Drug: Rituximab; Drug: Vincristine
- Phase 2: Alisertib (Experimental): Phase 2: Alisertib (MLN8237) at the Recommended Phase 2 Dose, ECT orally twice/day on Days 1-7 & rituximab as an IV infusion on Day 1 & vincristine IV on Days 1 & 8 in a 21 Day cycle for up to 8 cycles was planned but not conducted.
  Interventions: Drug: Alisertib (MLN8237); Drug: Rituximab; Drug: Vincristine

INTERVENTIONS:
Drug: Alisertib (MLN8237) — Alisertib (MLN8237) enteric coated tablet (ECT).
Drug: Rituximab — Rituximab IV infusion.
Drug: Vincristine — Vincristine IV Infusion.
  Arms: Dose Escalation, Alisertib 30 mg; Dose Escalation, Alisertib 40 mg; Dose Escalation, Alisertib 50 mg; Phase 2: Alisertib

SUMMARY:
This is a single-arm, open-label, multicenter, dose escalation, phase 1-2 study of alisertib (MLN8237) administered in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL)/transformed follicular lymphoma (TFL) treated with rituximab and vincristine. The study has three parts as follows:

Phase 1, Part 1: Safety lead-in cohort to evaluate alisertib (MLN8237) and rituximab.

Phase 1, Part 2: Dose escalation cohort to evaluate alisertib (MLN8237) + Rituximab + Vincristine and determine Phase 2 dose. Patients with other types of B-cell lymphoma (including mantle cell or Burkitt's lymphoma may enroll in Parts 1 and 2.

Phase 2: Alisertib (MLN8237) + Rituximab + Vincristine in patients with relapsed or refractory DLBCL or TFL at recommended Phase 2 dose.

Note that in 2013 Sponsor decision was taken to not initiate the phase 2 portion of the trial, which would have investigated the triplet at the recommended phase 2 dose identified in part 2. This decision was based on reprioritization within the company and not on any clinical or safety outcomes observed.

DETAILED DESCRIPTION:
The drug tested in this study was called alisertib. Alisertib was tested to treat people who have relapsed or refractory diffuse large B-cell lymphoma or other aggressive B-cell lymphomas. This study looked at safety, any anti-tumor effect, and it also determined a recommended dose of alisertib plus rituximab and alisertib plus rituximab and vincristine to take into further studies. Pharmacokinetic blood samples were studied to characterize any effects on the concentration of each of the drugs when administered together .

The study enrolled 45 patients. Participants received the following treatments:

Phase 1

* Alisertib 50 mg + rituximab in the Safety Lead-in
* Alisertib 30 mg + rituximab + vincristine in the Dose Escalation
* Alisertib 40 mg + rituximab + vincristine in the Dose Escalation
* Alisertib 50 mg + rituximab + vincristine in the Dose Escalation

All participants were asked to take one alisertib table twice a day for 7 days in each cycle for up to 8 cycles along with rituximab on Day 1 of each cycle; some patients also received vincristine on Day 1 and Day 8 of each cycle. All participants with documented disease response or stabilization could continue with alisertib single-agent therapy for an additional 2 years or more.

This multi-center trial was conducted in the USA. The overall time to participate in this study was up to 5.2 years. Participants made multiple visits to the clinic, plus a final visit 30 days after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL)/transformed follicular lymphoma (TFL). Note: Patients with Mantle Cell or Burkitt's lymphoma may be eligible for enrollment to the safety lead-in and dose escalation cohorts, parts 1 & 2 only
* Relapsed or refractory after at least 1 prior systemic treatment for aggressive lymphoma (including anthracycline unless contra-indicated). Relapse following an autologous stem cell transplant is allowed.
* Relapsed after autologous stem cell transplantation or not be eligible for autologous stem cell transplantation or refuse autologous stem cell transplantation. Patients enrolled to the phase 2 part must have received prior rituximab.
* Measurable disease as specified in study protocol
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Female patients who are post menopausal for at least 1 year, surgically sterile, or agree to practice 2 effective methods of contraception through 30 days after the last dose of alisertib (MLN8237) or agree to abstain from heterosexual intercourse. Patients should also use effective contraception for 12 months following the last dose of rituximab and 1 month following the last dose of alisertib (MLN8237.
* Male patients who agree to practice effective barrier contraception through 4 months after the last dose of MLN8237 or agree to abstain from heterosexual intercourse
* Voluntary written consent

Exclusion Criteria

* Received more than 4 prior systemic treatment regimens for lymphoma
* Known human immunodeficiency virus (HIV) positive or acquired immunodeficiency syndrome (AIDS)-related illness; hepatitis B virus, or hepatitis C virus; known history of Charcot-Marie-Tooth disease or polio
* Autologous stem cell transplant less than 3 months prior to enrollment
* Patients who have undergone allogeneic stem cell or organ transplantation any time
* Systemic antineoplastic therapy, including glucocorticoids or treatment with an investigational agent within 14 days preceding the first dose of study drug treatment. Steroids are permitted for administration with rituximab to prevent or treat infusion reaction
* Treatment with nitrosoureas, mitomycin C, rituximab, alemtuzumab, or other unconjugated antibody treatment within 42 days (21 days if clear evidence of progressive disease) prior to the first day of study drug treatment
* Treatment with radioimmunoconjugates or toxin immunoconjugates, such as ibritumomab-tiuxetan, or tositumomab, within 12 weeks prior to the first day of study drug treatment
* Radiotherapy within 21 days prior to the first dose of study drug treatment
* Treatment with enzyme-inducing antiepileptic drugs, such as phenytoin, carbamazepine, or phenobarbital, or with rifampin, rifabutin, rifapentine, or St. John's wort, within 14 days prior to the first dose of alisertib (MLN8237) also not permitted during study
* Cardiac status as described in protocol
* Major surgery, serious infection, or infection requiring systemic antibiotic therapy within 14 days prior to the first dose of study treatment
* History of hemorrhagic or thrombotic cerebrovascular event in the past 12 months
* Clinically uncontrolled central nervous system involvement
* Inability to receive IV rituximab or vincristine, or to swallow tablets or inability or unwillingness to avoid taking anything by mouth except for water and prescribed medications for 2 hours before and 1 hour after each dose of alisertib (MLN8237)
* History of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness
* Female patients who are lactating or pregnant
* Serious medical or psychiatric illness or laboratory abnormality that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol
* Clinically apparent ≥ Grade 2 neuropathy due to any cause in the 3 months prior to enrollment, or history of ≥ Grade 3 neuropathy related to vincristine at any time
* Prior treatment with Aurora A-targeted agents, including alisertib (MLN8237)
* Patients who have received myeloid growth factors or platelet transfusion within 14 days prior to the first dose of study treatment
* Patients with known hypersensitivity to rituximab, vincristine (or vinca alkaloids), or their diluents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-08-09 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2016-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (25):
- United States (15):
  - Tucson, Arizona
  - Beverly Hills, California
  - Burbank, California
  - Miami, Florida
  - Lexington, Kentucky
  - Worcester, Massachusetts
  - New York, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania
  - Germantown, Tennessee
  - Memphis, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Burlington, Vermont
- Italy (4):
  - Orbassano, Torino
  - Genova
  - Palermo
  - Roma
- Spain (2):
  - Madrid
  - Seville
- United Kingdom (4):
  - Aberdeen, Grampian Region
  - London, Greater London
  - Southampton, Hampshire
  - Birmingham, West Midlands

REFERENCES:
- [Derived] Kelly KR, Friedberg JW, Park SI, McDonagh K, Hayslip J, Persky D, Ruan J, Puvvada S, Rosen P, Iyer SP, Stefanovic A, Bernstein SH, Weitman S, Karnad A, Monohan G, VanderWalde A, Mena R, Schmelz M, Spier C, Groshen S, Venkatakrishnan K, Zhou X, Sheldon-Waniga E, Leonard EJ, Mahadevan D. Phase I Study of the Investigational Aurora A Kinase Inhibitor Alisertib plus Rituximab or Rituximab/Vincristine in Relapsed/Refractory Aggressive B-cell Lymphoma. Clin Cancer Res. 2018 Dec 15;24(24):6150-6159. doi: 10.1158/1078-0432.CCR-18-0286. Epub 2018 Aug 6. PMID 30082475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the Phase 1 portion of the study at 10 investigative sites in the United States from 09 August 2011 to 05 October 2016. The Phase 2 portion of the study was cancelled by the sponsor.
Pre-assignment Details: Participants with a diagnosis of relapsed or refractory Diffuse Large B-cell lymphoma (DLBCL)/transformed Follicular lymphoma (TFL), Mantle Cell lymphoma, or Burkitt's Lymphoma were enrolled to receive alisertib open label at doses 30 mg, 40 mg or 50 mg.
Groups:
- Dose Escalation, Alisertib 30 mg: Alisertib 30 mg, ECT, orally, BID, on Days 1 to 7 followed by a 14-day rest period plus rituximab 375 mg/m^2, IV, infusion on Day 1, plus vincristine 1.4 mg/m^2, IV (max 2 mg), on Days 1 and 8 in a 21-day cycle for up to 8 cycles. Following 8 cycles of treatment (or early discontinuation of rituximab and/or vincristine) all participants with documented disease response or stabilization may continue with alisertib single-agent therapy for up to 2 years.
- Dose Escalation, Alisertib 40 mg: Alisertib 40 mg, ECT, orally, BID, on Days 1 to 7 followed by a 14-day rest period plus rituximab 375 mg/m^2, IV, infusion on Day 1 plus vincristine 1.4 mg/m^2, IV (max 2 mg), on Days 1 and 8 in a 21-day cycle for up to 8 cycles. Following 8 cycles of treatment (or early discontinuation of rituximab and/or vincristine) all participants with documented disease response or stabilization may continue with alisertib single-agent therapy for up to 2 years.
- Dose Escalation, Alisertib 50 mg: Alisertib 50 mg, ECT, orally, BID, on Days 1 to 7 followed by a 14-day rest period plus rituximab 375 mg/m^2, IV, infusion on Day 1 plus vincristine 1.4 mg/m^2, IV (max 2 mg), on Days 1 and 8 in a 21-day cycle for up to 8 cycles. Following 8 cycles of treatment (or early discontinuation of rituximab and/or vincristine) all participants with documented disease response or stabilization may continue with alisertib single-agent therapy for up to 2 years.
Period: Overall Study
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg | Phase 2: Alisertib
Started | 13 | 4 | 25 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 13 | 4 | 25 | 3 | 0
Not completed — Progressive Disease | 10 | 3 | 11 | 1 | 0
Not completed — Symptomatic Deterioration | 2 | 0 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 5 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population was defined as all participants who receive any amount of alisertib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg | Total
Number analyzed (Participants) | 13 | 4 | 25 | 3 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (14.06) | 51.3 (21.65) | 62.8 (10.51) | 66.7 (12.86) | 61.3 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 10 | 2 | 16
  Male | 10 | 3 | 15 | 1 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 7 | 1 | 6 | 1 | 15
  Not Hispanic or Latino | 6 | 3 | 19 | 2 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12 | 4 | 21 | 3 | 40
  Black or African American | 0 | 0 | 2 | 0 | 2
  Asian | 1 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 1 | 0 | 1
  Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 4 | 25 | 3 | 45
Height [Mean (Standard Deviation); unit: cm] | 167.9 (10.90) | 178.2 (7.15) | 168.4 (10.76) | 166.5 (5.32) | 169.0 (10.44)
Weight [Mean (Standard Deviation); unit: kg] | 70.98 (16.18) | 89.51 (23.89) | 82.21 (16.4) | 71.94 (14.55) | 78.93 (17.46)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body surface area (m^²)=square root [height (cm)×weight (kg)/3600].
  m^2 | 1.815 (0.25) | 2.093 (0.31) | 1.940 (0.23) | 1.823 (0.21) | 1.910 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Vital Signs Findings (Treatment Related and Unrelated) [Phase 1]
Description: Vital sign parameters: blood pressure, heart rate and temperature determined by the investigator to be clinically significant were reported as adverse events.
Time Frame: First dose of alisertib through 30 days after the last dose of alisertib (Up to 5.2 Years)
Population: Safety Population was defined as all participants who receive any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 13 | 4 | 25 | 3
participants
  Hypotension | 0 | 0 | 3 | 1
  Orthostatic hypotension | 2 | 2 | 0 | 0
  Hypertension | 1 | 0 | 0 | 0
  Pyrexia | 3 | 0 | 2 | 1

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiograms (ECGs) [Phase 1]
Description: Abnormal ECGs findings determined by the investigator to be clinically significant were reported as adverse events.
Time Frame: First dose of alisertib through 30 days after the last dose of alisertib (Up to 5.2 Years)
Population: Safety Population was defined as all participants who receive any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 13 | 4 | 25 | 3
participants | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Multigated Acquisition (MUGA)/ Echocardiogram (ECHO) [Phase 1]
Description: Abnormal changes in MUGA and ECHO findings determined by the investigator to be clinically significant were reported as adverse events.
Time Frame: First dose of alisertib through 30 days after the last dose of alisertib (Up to 5.2 Years)
Population: Safety Population was defined as all participants who receive any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 13 | 4 | 25 | 3
participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination Findings [Phase 1]
Description: Abnormal Physical Examination findings determined by the investigator to be clinically significant were reported as Adverse Events.
Time Frame: First dose of alisertib through 30 days after the last dose of alisertib (Up to 5.2 Years)
Population: Safety Population was defined as all participants who receive any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 13 | 4 | 25 | 3
participants | 0 | 0 | 2 | 2

5. Primary Outcome: Number of Participants With Clinically Significant Laboratory Tests Reported as Adverse Events [Phase 1]
Description: Abnormal treatment-emergent Chemistry and Hematology Laboratory values determined by the investigator to be clinically significant were reported as adverse events.
Time Frame: First dose of alisertib through 30 days after the last dose of alisertib (Up to 5.2 Years)
Population: Safety Population was defined as all participants who receive any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 13 | 4 | 25 | 3
participants
  Anaemia | 6 | 3 | 14 | 2
  Neutropenia | 7 | 2 | 11 | 2
  Febrile neutropenia | 0 | 0 | 4 | 3
  Leukopenia | 8 | 2 | 9 | 3
  Lymphopenia | 2 | 2 | 1 | 1
  Thrombocytopenia | 7 | 1 | 7 | 3
  Hypokalaemia | 5 | 0 | 6 | 2
  Hyperkalaemia | 0 | 0 | 1 | 0
  Hypomagnesaemia | 2 | 0 | 5 | 1
  Hypermagnesaemia | 0 | 0 | 0 | 1
  Hypocalcaemia | 2 | 0 | 1 | 1
  Hypercalcaemia | 1 | 0 | 2 | 0
  Hyperglycaemia | 1 | 1 | 2 | 1
  Hypoalbuminaemia | 3 | 0 | 0 | 2
  Hyponatraemia | 2 | 0 | 0 | 1
  Hypernatraemia | 0 | 0 | 1 | 0
  Hypophosphataemia | 1 | 0 | 1 | 1
  Neutrophil count decreased | 1 | 0 | 3 | 1
  Lymphocyte count decreased | 1 | 0 | 0 | 0
  White blood cell count decreased | 0 | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 1 | 2
  Alanine aminotransferase increased | 0 | 0 | 0 | 2
  Blood bilirubin increased | 1 | 0 | 0 | 0
  Platelet count decreased | 1 | 0 | 1 | 1

6. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Phase 1]
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose of alisertib through 30 days after the last dose of alisertib (Up to 5.2 Years)
Population: Safety Population was defined as all participants who receive any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 13 | 4 | 25 | 3
participants | 13 | 4 | 25 | 3

7. Primary Outcome: Overall Response Rate [Phase 2]
Description: Overall Response Rate was defined as the percentage of participants with Complete Response (CR) or Partial Response (PR) as assessed by the investigator using International Working Group (IWG) Criteria. CR is defined as the disappearance of all evidence of disease and PR is defined as regression of measurable disease and no new sites.
Time Frame: At the end of Cycle 2, at the end of every second treatment cycle until 6 months, then every 12 weeks thereafter, approximately 2 years
Population: The Phase 2 portion of the study was cancelled by the sponsor.
Arm/Group | Phase 2: Alisertib
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Response Rate as Assessed by the Investigator [Phase 1]
Description: as for outcome 7
Time Frame: First dose of alisertib through 30 days after the last dose of alisertib (Up to 5.2 Years)
Population: Response-Evaluable Population was defined as all participants with measurable disease who received at least 1 dose of alisertib and had at least 1 post-baseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 12 | 3 | 20 | 2
percentage of participants | 25 [5 to 57] | 33 [0.84 to 91] | 45 [23 to 68] | 50 [1 to 99]

9. Secondary Outcome: Complete Response Rate [Phase 2]
Description: Complete response rate was defined as the percentage of participants with Complete Response (CR). CR was assessed by the investigator using International Working Group (IWG) Criteria. CR is defined as the disappearance of all evidence of disease.
Time Frame: Duration of study until disease progression, approximately 2 years
Population: Phase 2 portion of the study was cancelled by the sponsor.
Arm/Group | Phase 2: Alisertib
Number analyzed (Participants) | 0

10. Secondary Outcome: Duration of Response (DOR) [Phase 2]
Description: DOR was defined as the time from the date of first documentation of a response to the date of first documentation of Progressive Disease (PD).
Time Frame: Duration of study until disease progression, approximately 2 years
Population: Phase 2 portion of the study was cancelled by the sponsor.
Arm/Group | Phase 2: Alisertib
Number analyzed (Participants) | 0

11. Secondary Outcome: Progression Free Survival (PFS) [Phase 2]
Description: PFS was defined as the time from the date of first study drug administration to the date of first documentation of PD or death.
Time Frame: Duration of study until disease progression, approximately 2 years
Population: The Phase 2 portion of the study was cancelled by the sponsor.
Arm/Group | Phase 2: Alisertib
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Phase 2]
Description: as for outcome 6
Time Frame: From screening period to 30 days after last dose of study drug, approximately 2 years
Population: Phase 2 portion of the study was cancelled by the sponsor.
Arm/Group | Phase 2: Alisertib
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Findings [Phase 2]
Description: as for outcome 1
Time Frame: From screening period to 30 days after last dose of study drug, approximately 2 years
Population: Phase 2 portion of the study was cancelled by the sponsor.
Arm/Group | Phase 2: Alisertib
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiograms (ECGs) [Phase 2]
Time Frame: From screening period to 30 days after last dose of study drug, approximately 2 years
Population: Phase 2 portion of the study was cancelled by the sponsor.
Arm/Group | Phase 2: Alisertib
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Changes in Multigated Acquisition (MUGA)/ Echocardiogram (ECHO) [Phase 2]
Time Frame: From screening period to 30 days after last dose of study drug, approximately 2 years
Population: Phase 2 portion of the study was cancelled by the sponsor.
Arm/Group | Phase 2: Alisertib
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Tests Reported as Adverse Events [Phase 2]
Time Frame: From screening period to 30 days after last dose of study drug, approximately 2 years
Population: Phase 2 portion of the study was cancelled by the sponsor.
Arm/Group | Phase 2: Alisertib
Number analyzed (Participants) | 0

17. Secondary Outcome: Cmax: Maximum Plasma Concentration for Alisertib
Time Frame: Cycle 1 Days 1 and 7 prior to morning alisertib dose and multiple time-points (up to 12 hours) post-dose
Population: Alisertib Pharmacokinetic (PK)-Evaluable Population was defined as all participants with sufficient dosing and alisertib concentration-time data to permit non-compartmental PK analysis. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: nanoMolar (nM)
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 13 | 4 | 25 | 3
nanoMolar (nM)
  Day 1 | 1624.1 (929.68) | 893.3 (350.03) | 1159.7 (391.78) | 1746.7 (594.75)
  Day 7: number analyzed (Participants) | 12 | 4 | 20 | 2
  Day 7 | 2915.8 (1537.03) | 1672.5 (183.92) | 2223.3 (1217.22) | 3670.0 (1541.49)

18. Secondary Outcome: Tmax: Time to First Occurrence of Cmax fo Alisertib
Time Frame: Cycle 1 Days 1 and 7 prior to morning alisertib dose and multiple time-points (up to 12 hours) post-dose
Population: Alisertib PK-Evaluable Population was defined as all participants with sufficient dosing and alisertib concentration-time data to permit non-compartmental PK analysis. Number analyzed is the number of participants with data available at the given time-point.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 13 | 4 | 25 | 3
hours (hr)
  Day 1 | 3.0 [2 to 8] | 3.5 [3 to 6] | 3.0 [1 to 12] | 6.1 [3 to 12]
  Day 7: number analyzed (Participants) | 12 | 4 | 20 | 2
  Day 7 | 2.0 [0 to 8] | 3.1 [2 to 6] | 3.1 [2 to 8] | 2.5 [2 to 3]

19. Secondary Outcome: AUCt: Area Under the Concentration Time Curve Over the Dosing Interval From Time 0 to Time t for Alisertib
Time Frame: Cycle 1 Days 1 and 7 prior to morning alisertib dose and multiple time-points (up to 12 hours) post-dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: nanomoles/liter*hour (nmol/L*hr)
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 13 | 4 | 25 | 3
nanomoles/liter*hour (nmol/L*hr)
  Day 1: number analyzed (Participants) | 12 | 4 | 22 | 3
  Day 1 | 10116.7 (6683.97) | 5817.5 (2966.26) | 8005.9 (3251.32) | 13096.7 (7453.39)
  Day 7: number analyzed (Participants) | 12 | 4 | 20 | 2
  Day 7 | 21812.5 (13090.21) | 12227.5 (3480.09) | 17996.0 (11555.15) | 33800.0 (16263.46)

20. Secondary Outcome: Cmax: Maximum Plasma Concentration for Vincristine
Time Frame: Cycles 1 and 2 on Day 1 prior to injection of vincristine and multiple time-points (up to 72 hours) post-dose
Population: Vincristine PK-evaluable population was defined as all participants with sufficient dosing and vincristine concentration-time data to permit non-compartmental PK analysis. Safety Lead-in arm did not receive vincristine. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 4 | 25 | 3
ng/mL
  Cycle 1, Day 1 | 132.2 (54.57) | 105.4 (78.93) | 158.4 (67.94)
  Cycle 2, Day 1: number analyzed (Participants) | 4 | 17 | 2
  Cycle 2, Day 1 | 113.9 (53.86) | 124.4 (157.70) | 122.3 (36.42)

21. Secondary Outcome: AUCt: Area Under the Concentration-time Time Curve Over the Dosing Interval From Time 0 to Time t for Vincristine
Time Frame: Cycles 1 and 2 on Day 1 prior to injection of vincristine and multiple time-points (up to 72 hours) post-dose
Population: Vincristine PK-evaluable population was defined as all participants with sufficient dosing and vincristine concentration-time data to permit non-compartmental PK analysis. Safety Lead-in arm did not receive vincristine Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Arm/Group | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 4 | 24 | 3
ng/mL*hr
  Cycle 1, Day 1 | 69.8 (9.92) | 69.1 (33.24) | 104.1 (43.34)
  Cycle 2, Day 1: number analyzed (Participants) | 2 | 17 | 2
  Cycle 2, Day 1 | 60.8 (2.26) | 72.8 (30.40) | 72.2 (32.60)

22. Secondary Outcome: AUC∞: Area Under the Concentration-time Curve From Time 0 to Infinity for Vincristine
Time Frame: Cycles 1 and 2 on Day 1 prior to injection of vincristine and multiple time-points (up to 72 hours) post-dose
Population: Vincristine PK-evaluable population was defined as participants with sufficient dosing and concentration-time data to permit non-compartmental PK analysis. Safety Lead-in arm did not receive vincristine. Number analyzed is the number of participants with data available at the time-point. No data was collected for the alisertib 50 mg arm in Cycle 2.
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Arm/Group | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 4 | 22 | 3
ng/mL*hr
  Cycle 1, Day 1 | 77.9 (11.25) | 84.8 (36.21) | 116.8 (44.95)
  Cycle 2, Day 1: number analyzed (Participants) | 3 | 16 | 0
  Cycle 2, Day 1 | 69.0 (4.45) | 82.7 (35.39) |

23. Secondary Outcome: T1/2: Terminal Disposition Phase Half-life for Vincristine
Time Frame: Cycles 1 and 2 on Day prior to injection of vincristine and multiple time-points (up to 72 hours) post-dose
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Number analyzed (Participants) | 4 | 25 | 3
nanogram/milliliter (ng/mL)
  Cycle 1, Day 1: number analyzed (Participants) | 4 | 22 | 3
  Cycle 1, Day 1 | 20.2 (5.04) | 20.0 (5.89) | 25.6 (4.55)
  Cycle 2, Day 1: number analyzed (Participants) | 3 | 16 | 0
  Cycle 2, Day 1 | 19.9 (0.92) | 20.2 (4.66) |

ADVERSE EVENTS:
Time Frame: First dose of alisertib through 30 days after the last dose of alisertib (Up to 5.2 Years)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Safety Lead-in | Dose Escalation, Alisertib 30 mg | Dose Escalation, Alisertib 40 mg | Dose Escalation, Alisertib 50 mg
Serious Adverse Events (participants affected / at risk) | 6/13 | 1/4 | 12/25 | 3/3
Other Adverse Events (participants affected / at risk) | 13/13 | 4/4 | 25/25 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Lead-in (N=13) | Dose Escalation, Alisertib 30 mg (N=4) | Dose Escalation, Alisertib 40 mg (N=25) | Dose Escalation, Alisertib 50 mg (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with alisertib 40 mg BID and is not related.
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 — Two treatment-emergent deaths occurred during treatment with alisertib 50 mg BID and alisertib 40 mg BID and are not related.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with 50 mg BID and is not related.
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Lead-in (N=13) | Dose Escalation, Alisertib 30 mg (N=4) | Dose Escalation, Alisertib 40 mg (N=25) | Dose Escalation, Alisertib 50 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 15 | 2
Leukopenia (Blood and lymphatic system disorders) | 8 | 2 | 9 | 3
Neutropenia (Blood and lymphatic system disorders) | 7 | 2 | 11 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 1 | 8 | 3
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 16 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 14 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 9 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 6 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 11 | 2
Chills (General disorders) | 2 | 0 | 3 | 0
Oedema peripheral (General disorders) | 1 | 1 | 3 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1
Early satiety (General disorders) | 0 | 0 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0
Infusion site erythema (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Temperature regulation disorder (General disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 7 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 6 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 5 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 6 | 1
Headache (Nervous system disorders) | 1 | 1 | 5 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 4 | 1
Somnolence (Nervous system disorders) | 5 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Tongue paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Platelet count decreased (Investigations) | 1 | 0 | 1 | 1
Weight decreased (Investigations) | 1 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 4 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hydroureter (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 2 | 0
Ocular icterus (Eye disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal ulceration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The Phase 2 portion of the study was cancelled by the sponsor; this was an administrative decision not based on any clinical or safety outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.